CLINICAL TRIAL: NCT01571401
Title: Trying Activity in Kidney Cancer Survivors (TRACKS) Trial: A Randomized Controlled Trial Comparing the Effects of Supervised Physical Activity Versus Supervised Physical Activity Plus Behavioural Counselling
Brief Title: Trying Activity in Kidney Cancer Survivors (TRACKS) Trial
Acronym: TRACKS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: TRACKS Trial for Kidney Cancer
Record Dates: First submitted 2012-04-02; First posted 2012-04-05 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2012-04

CONDITIONS: Supervised Physical Activity Plus Exercise Counseling; Supervised Physical Activity Plus Behavioural Counseling
Keywords: Kidney cancer survivors; Randomized Controlled Trial; Physical Activity; Theory of Planned Behaviour; Quality of life
MeSH Terms: conditions — Motor Activity | interventions — Clinical Trials as Topic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Supervised PA plus Exercise Counselling (Experimental): Participants will be provided with six individual supervised exercise sessions with a physical activity specialist that will taper to an unsupervised program by the end of the intervention. Over the 4-week period, this group will be required to attend two sessions per week for weeks 1-2, and one session per week for weeks 3-4 at fitness centre. In order to achieve the physical activity guidelines established by the current public health recommendations, additional unsupervised sessions will be prescribed. In addition to the supervised sessions, traditional exercise counselling will be provided to teach proper technique, how to monitor intensity, and to progress PA safely and effectively to achieve the public health physical activity guidelines
  Interventions: Behavioral: Trying Activity for Kidney Cancer Survivors (TRACKS) Trial
- Supervised PA plus behavioural counselling (Experimental): In addition to the same supervised PA sessions as the SPA group, participants in this group will receive six individual "face-to-face" behavioural counselling sessions with a physical activity specialist. These counselling sessions will be combined with the supervised PA sessions, and will be provided directly following the supervised PA session. Counselling strategies will be based on the TPB and will target the unique benefits of PA for kidney cancer survivors, strategies for making PA enjoyable, for overcoming barriers, for including social support from family and friends, time management, self-monitoring, goal setting, and planning.
  Interventions: Behavioral: Trying Activity for Kidney Cancer Survivors (TRACKS) Trial

INTERVENTIONS:
Behavioral: Trying Activity for Kidney Cancer Survivors (TRACKS) Trial — Participants in both arms will be provided with six individual supervised exercise sessions with a physical activity specialist that will taper to an unsupervised program by the end of the intervention. Over the 4-week period, both groups will be required to attend two sessions per week for weeks 1-2, and one session per week for weeks 3-4 at the Behavioural Medicine Fitness Centre at the University of Alberta. In order to achieve the PA guidelines established by the current public health recommendations, additional unsupervised sessions will be prescribed.

SUMMARY:
Objectives: The purpose of this study is to find out if a new program can help kidney cancer survivors (KCS) increase their physical activity (PA) and improve their quality of life (QoL).

Methods: Fifty KCS will be recruited from a previous study using the Alberta Cancer Registry. Participants will undergo submaximal exercise testing, a physical function test and measures of height and weight, which will be completed at baseline and the end of the physical activity program (at 12 weeks). Participants will also complete questionnaires on PA and QoL at the baseline, after the supervised portion of the program (at 4 weeks), and at the end of the entire program (at 12 weeks). Following baseline assessments, participants will be randomly assigned to either: (1) supervised physical activity plus traditional exercise counseling or (2) supervised physical activity plus behavioural counseling. Participants will be asked to attend six individual supervised exercise and counseling sessions over a 4-week period with a PA specialist that eventually tapers to a home-based program by the end of the program.

Implications: The investigators hope that this PA intervention for KCS is feasible and results in meaningful improvements in health outcomes that can be translated to public health practice.

DETAILED DESCRIPTION:
Background: Despite the reported benefits of physical activity (PA), the majority of cancer survivors are not meeting public health PA guidelines. Most PA intervention studies have used supervised exercise and demonstrated benefits. However, these studies have also found that PA declines significantly after the supervised intervention is completed. Consequently, interventions are needed to ensure longer term adherence after short term supervised exercise interventions. Although several of behaviour change interventions have supported positive increases in PA, no study to date has examined the effects of adding behavioural counseling to a standard supervised exercise program and no study has focused on kidney cancer survivors (KCS).

Objectives: The primary purpose of the Trying Activity in Kidney Cancer Survivors (TRACKS) Trial is to compare the effects of a supervised physical activity program plus traditional exercise counseling (SPA) versus a supervised physical activity plus motivationally-enhanced behavioural counseling (SPA+BC) on change in self-reported moderate/vigorous PA between baseline, post-intervention, and 12-week follow-up among KCS. The secondary outcomes are changes in self-reported quality of life (QoL), body composition (anthropometric measures), cardiorespiratory fitness, physical function, and motivational constructs from the Theory of Planned Behaviour (TPB) constructs.

Methods: The study will pilot a two-armed, randomized controlled trial of 50 KCS. KCS will be recruited from a previous study using the Alberta Cancer Registry. Eligibility will include: a) between 18-80 years of age, b) diagnosed with Stage I-IIIa kidney cancer, and g) interested in increasing their physical activity. Following the screening procedure and prior to randomization, participants will undergo submaximal exercise testing on a treadmill to ensure that they are able to exercise safely at a moderate-to-vigorous intensity. Randomization will occur after all baseline measurements have been completed. The goal of the intervention, based on current public health recommendations, will be to gradually increase all participants by at least 60 minutes of moderate intensity PA or 30 minutes of vigorous intensity PA to a minimum of 150 minutes of moderate intensity PA or 75 minutes of vigorous intensity PA per week. Participants in both arms will be provided with six individual supervised exercise sessions with a physical activity specialist that will taper to an unsupervised program by the end of the intervention. Participants assigned to the SPA group will be given an individualized prescription at a moderate-to-vigorous intensity. They will also receive traditional exercise counseling to teach proper PA technique, how to monitor intensity, and to progress PA safely and effectively to achieve the public health PA guidelines. For the SPA+BC group, participants will receive the same supervised PA sessions with the addition of six individual "face-to-face" behavioural counseling sessions with a physical activity specialist. These behaviour counseling sessions will include training in behavioural strategies to promote the adoption and long-term maintenance of PA. Measurements for the primary and secondary endpoints will be assessed at baseline (pre-intervention), 4 weeks (post-intervention), and 12 weeks follow-up.

Conclusion: The study results can be used to determine if a behavior change intervention for KCS based on the TPB results in potentially meaningful improvements in PA and selected health outcomes.

ELIGIBILITY:
Inclusion Criteria:

Screening evaluations will be conducted on interested participants and eligibility criteria include the following: a) between the ages of 18 to 80 years of age, histologically confirmed kidney cancer (Stage I-IIIa); b) ability and willingness to effectively communicate with the study coordinator and complete all questionnaires involved in the study in English; c) able to attend the supervised PA sessions and not planning to be away for three consecutive days for the duration of the program; and d) interested in increasing their PA by at least 60 minutes of moderate PA or 30 minutes of vigorous PA. Following the screening procedure and prior to randomization, consenting participants that are deemed eligible will undergo submaximal exercise testing to ensure that they are able to exercise safely at a moderate-to-vigorous intensity. Two stages of the treadmill test must be successfully completed with acceptable heart rate and blood pressure responses before any remaining baseline tests will be conducted including a physical function test, anthropometric testing, and PA behaviour, quality of life, and determinants questionnaire.

Exclusion Criteria:

The researchers can remove the participants from the study early for reasons such as a cancer recurrence, doctor feels that the participant is unable to participate in a physical activity program and/or participate in the follow up fitness testing, and/or two stages of the treadmill test cannot be completed.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
self-reported moderate/vigorous physical activity | 12 weeks
  A modified version of the validated Leisure Score Index (LSI) from the Godin Leisure-Time Exercise Questionnaire (GLTEQ), that has been extensively validated, will be used to assess PA behavior. Participants will be asked to recall their average weekly frequency and duration of light (minimal effort, no perspiration), moderate (not exhausting, light perspiration), and vigorous (heart beats rapidly, sweating) PA that lasted at least 10 minutes and was done during free time in the past month.

SECONDARY OUTCOMES:
Quality of life (QoL) | 12 weeks
  Disease-specific QoL will be assessed by the well-validated Functional Assessment of Cancer Therapy-Fatigue (FACT-F) scale which includes the 27 items from the FACT-General (FACT-G) scale plus the 13 item fatigue subscale.
  Generic QoL will also be assessed using the RAND (Research and Development)-36 Health Status Inventory, which contains 36 items that yield eight health domains with multi-item scales.
Theory of Planned Behaviour (TPB) | 12 weeks
  TPB items will be assessed by asking questions related to instrumental and affective attitude, descriptive and injunctive norms, perceived behavioural control, intention, and planning using a likert-type response format.
Anthropometric measures | 12 weeks
  Measurements of height, weight, and circumferences will be used to estimate body composition. Height will be measured using a stadiometer to the nearest 0.1 cm. Weight will be measured using a balance beam scale to the nearest 0.1 kg. Height and weight will be used to calculate body mass index (BMI) [weight per height squared (kg/m²)].
cardiorespiratory fitness | 12 weeks
  Participants will undergo sub-maximal aerobic testing to assess aerobic fitness and estimate VO2max from simple heart rate measurements. The test used will be a modified Balke Test performed on a treadmill to 85% of their maximal heart rate or exhaustion.
physical function | 12 weeks
  The Seniors' Fitness Test (SFT) will be used to assess physical fitness/function in older adults aged 60 to 90+ years old. The SFT consists of a battery of six assessment items used to determine mobility-related fitness parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Trinh, MA, Principal Investigator — University of Alberta
Locations (1):
- Behavioural Medicine Fitness Centre, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Trinh L, Plotnikoff RC, Rhodes RE, North S, Courneya KS. Associations between physical activity and quality of life in a population-based sample of kidney cancer survivors. Cancer Epidemiol Biomarkers Prev. 2011 May;20(5):859-68. doi: 10.1158/1055-9965.EPI-10-1319. Epub 2011 Apr 5. PMID 21467240
- [Background] Trinh L, Plotnikoff RC, Rhodes RE, North S, Courneya KS. Physical activity preferences in a population-based sample of kidney cancer survivors. Support Care Cancer. 2012 Aug;20(8):1709-17. doi: 10.1007/s00520-011-1264-z. Epub 2011 Sep 24. PMID 21947412